CLINICAL TRIAL: NCT03313778
Title: A Phase 1, Open-Label, Multicenter Study to Assess the Safety, Tolerability, and Immunogenicity of mRNA-4157 Alone and in Combination in Participants With Solid Tumors
Brief Title: Safety, Tolerability, and Immunogenicity of mRNA-4157 Alone and in Combination in Participants With Solid Tumors
Acronym: KEYNOTE-603
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: mRNA-4157-P101; 2023-505192-77-00 (Other: EU CT Number)
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumors
Keywords: mRNA-4157; PCV; pembrolizumab; Moderna; intismeran autogene
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part A: Dose Escalation and Dose Expansion (Experimental): Participants will receive mRNA-4157 via an intramuscular (IM) injection on Day 1 of each 21-day cycle for up to 9 cycles.
  Interventions: Biological: mRNA-4157
- Part B: Dose Escalation and Dose Expansion (Experimental): Participants will receive mRNA-4157 via an IM injection on Day 1 of each 21-day cycle for up to 9 cycles and pembrolizumab via IV infusion on Day 1 of each 21-day cycle until progression, unacceptable toxicity, or up to 35 cycles (approximately 2 years of treatment), whichever is sooner.
  Interventions: Biological: mRNA-4157; Biological: Pembrolizumab
- Part A2: Dose Expansion (Experimental): Participants will receive mRNA-4157 via an IM injection on Day 1 of each 21-day cycle and a SoC treatment every 2 weeks (Q2W) on Day 1 of each 21-day cycle starting from Cycle 5 of mRNA-4157 for up to 12 cycles.
  Interventions: Biological: mRNA-4157; Biological: SoC Treatment
- Part C: Dose Expansion (Experimental): Participants will receive mRNA-4157 via IM injection on Day 1 of each 21-day cycle for up to 9 cycles and pembrolizumab via IV infusion on Day 1 of each 21-day cycle until progression, unacceptable toxicity, or up to 35 cycles (approximately 2 years of treatment), whichever is sooner.
  Interventions: Biological: mRNA-4157; Biological: Pembrolizumab
- Part D: Dose Expansion (Experimental): Participants will receive mRNA-4157 via IM injection on Day 1 of each 21-day cycle for up to 9 cycles and pembrolizumab via IV infusion on Day 1 of each 21-day cycle until progression, unacceptable toxicity, or up to 18 cycles (approximately 1 year of treatment), whichever is sooner.
  Interventions: Biological: mRNA-4157; Biological: Pembrolizumab
- Part E1: Dose Expansion (Experimental): Participants will receive mRNA-4157 via IM injection on Day 1 of each 21-day cycle, pembrolizumab every 6 weeks (Q6W) via IV infusion, and SoC chemotherapy every 3 weeks (Q3W) for up to 4 cycles during the perioperative and adjuvant phases.
  Interventions: Biological: mRNA-4157; Biological: Pembrolizumab; Biological: SoC Treatment
- Part E2: Dose Expansion (Experimental): Participants will receive mRNA-4157 via IM injection on Day 1 of each 21-day cycle, pembrolizumab Q6W via IV infusion, and SoC chemotherapy Q3W for up to 4 cycles during the perioperative and adjuvant phases.
  Interventions: Biological: mRNA-4157; Biological: Pembrolizumab; Biological: SoC Treatment
- Part E3: Dose Expansion (Experimental): Participants will receive mRNA-4157 via IM injection on Day 1 of each 21-day cycle, pembrolizumab Q3W via IV infusion, and SoC chemotherapy Q2W or Q3W for up to 4 cycles during the perioperative and adjuvant phases.
  Interventions: Biological: mRNA-4157; Biological: Pembrolizumab; Biological: SoC Treatment

INTERVENTIONS:
Biological: mRNA-4157 — IM injection
Biological: Pembrolizumab — Intravenous infusion
  Arms: Part B: Dose Escalation and Dose Expansion; Part C: Dose Expansion; Part D: Dose Expansion; Part E1: Dose Expansion; Part E2: Dose Expansion; Part E3: Dose Expansion
Biological: SoC Treatment — Intravenous infusion
  Other Names: Standard of care chemotherapy
  Arms: Part A2: Dose Expansion; Part E1: Dose Expansion; Part E2: Dose Expansion; Part E3: Dose Expansion

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and immunogenicity of mRNA-4157 alone and in combination in participants with solid tumors.

DETAILED DESCRIPTION:
This is a multi-part, dose-escalation study of mRNA-4157 monotherapy in participants with resected solid tumors (Part A), mRNA-4157 monotherapy lead-in and then in combination with standard of care (SoC) adjuvant chemotherapy followed by mRNA-4157 monotherapy in participants with resected pancreatic ductal adenocarcinoma (PDAC) (Part A2), mRNA-4157 in combination with pembrolizumab in participants with both unresectable (locally advanced or metastatic) solid tumors (Parts B and C) and adjuvant resected cutaneous melanoma (Part D), and mRNA-4157 in combination with pembrolizumab and SoC chemotherapy in peri-operative setting in participants with non-squamous non-small cell lung cancer (NSCLC) (Part E1), squamous cell NSCLC (Part E2), and gastric/ gastroesophageal (GEJ) cancer (Part E3). Parts A and B will include a dose escalation phase of the study to identify doses of mRNA-4157 for the expansion phase of the study. Doses of mRNA-4157 will be administered to participants in a dose escalation regimen. Participants in Parts A2, B, C, D, E1, E2 and E3 dose expansion phase will receive mRNA-4157 at a recommended dose for expansion.

ELIGIBILITY:
Inclusion Criteria:

* Parts A, A2, and D: Participants must be clinically disease-free at study entry (that is, participants in the adjuvant setting).
* Part B: Participants must have one of the histologically- or cytologically-confirmed unresectable (locally advanced or metastatic) protocol-specified solid malignancies, have measurable disease at study entry defined by RECIST 1.1., and be considered suitable for treatment with pembrolizumab; in this study pembrolizumab will be considered an investigational study drug.
* Part C: Participants must have one of the histologically- or cytologically confirmed unresectable (locally advanced or metastatic) protocol-specified solid malignancies, must not have received prior anti-programmed cell death protein 1 (PD-1)/programmed death -ligand 1 (PD-L1) therapy, and must have measurable disease at study entry defined by RECIST 1.1.
* Part A2: Participants with histologically confirmed PDAC who have undergone complete macroscopic resection(that is, R0 - no cancer cells within 1 mm of all resection margins or R1 - cancer cells present within 1 mm of one or more resection margins) who had no evidence of metastatic disease with adequate recovery from surgery to receive adjuvant therapy.
* Parts E1 and E2: Participants with untreated histologically/cytologically confirmed Stage II-IIIB NSCLC (per AJCC version 8) that is considered resectable of non-squamous (adenocarcinoma only) or squamous cell carcinoma histology, absence of major associated pathologies that increase the surgery risk to an unacceptable level, must have a tumor tissue sample available for NGS and PD-L1 IHC testing as defined in the Laboratory Manual.
* Part E3: Participants with untreated, locally advanced surgically resectable, histologically/cytologically confirmed, gastric/GEJ adenocarcinoma, as defined by a primary lesion that is T3 or greater or with the presence of any positive clinical nodes (N+) and without evidence of metastatic disease, measurable disease according to RECIST version 1.1, absence of major associated pathologies that increase the surgery risk to an unacceptable level, must have a tumor tissue sample available for NGS and PD-L1 IHC testing as defined in the Laboratory Manual.
* Part D: Participants with completely resected Stage II, III or IV cutaneous melanoma.
* Parts A, A2, and D: Participants must have a formalin-fixed paraffin embedded (FFPE) tumor sample available (for example, from their prior surgery) that is suitable for the next generation sequencing (NGS) required for this study.
* Parts B and C: Participants must have at least 1 lesion amenable to the mandatory fresh tumor biopsy at study entry.
* Participants must have resolution of toxic effect(s) (as specified in the protocol) from prior therapy to Grade 1 or less.
* Participant is willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study drug (male and female participants of childbearing potential), or for a specified time after the last dose of SoC chemotherapy per SoC product labeling, whichever is later.
* Participants with Performance Scale (PS) of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) PS.

Exclusion Criteria:

* Treatment with any of the following:

  1. Any investigational agents, anti-cancer monoclonal antibody, anti-cancer therapeutic vaccine, immunostimulant (for example, IL-2), or study drugs from a previous clinical study within 4 weeks of the first dose of mRNA-4157 or pembrolizumab (note only a 2 week wash out is required from prior pembrolizumab treatment)
  2. Any chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks of the first dose of mRNA-4157 or pembrolizumab
  3. Live-virus vaccination within 30 days of the first dose of mRNA-4157 or pembrolizumab. Seasonal flu vaccines that do not contain live virus are permitted.
  4. Any systemic steroid therapy or other form of immunosuppressive therapy within 7 days of the first dose of mRNA-4157 or pembrolizumab
  5. Transfusion of blood products (including platelets or red blood cells [RBCs]) or administration of colony stimulating factors (including granulocyte colony stimulating factor [G-CSF], granulocyte/macrophage colony stimulating factor [GM-CSF], or recombinant erythropoietin) within 1 week of the NGS blood sample during screening, and 4 weeks of the first dose of mRNA-4157 or pembrolizumab
* A history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating Investigator
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Previously identified hypersensitivity to chemotherapy agents that the participant would receive in their specific cohort or to components of the formulations used in this study
* Known additional malignancy that is progressing or requires active treatment, exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone curative therapy, or in situ cervical cancer.

Note: Additional inclusion/exclusion criteria may apply, per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2017-08-14 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Part A and A2: Baseline through 100 days after last mRNA-4157 dose; Parts B, C, D, E1, E2, and E3: Baseline through 90 days after last pembrolizumab dose

SECONDARY OUTCOMES:
Part C: Overall Response Rate (ORR): Number of Participants with Tumor Response (Partial or Complete) | Baseline through disease progression by Response Evaluation Criteria of Solid Tumors Version 1.1 (RECIST 1.1), start of new anti-cancer therapy, withdrawal of consent, death and last safety follow-up visit (up to approximately 3 years)
  ORR is defined as the proportion of participants whose best overall response is complete response (CR) or partial response (PR).
Part C: Duration of Response (DoR) | Baseline through disease progression by RECIST 1.1, start of new anti-cancer therapy, withdrawal of consent, death and last safety follow-up visit (up to approximately 3 years)
  DoR is defined as time from first tumor response (partial or complete) until either radiological disease progression, clinical/symptomatic disease progression or death (whichever is sooner).
Part C: Progression Free Survival (PFS) | Baseline through disease progression by RECIST 1.1, start of new anti-cancer therapy, withdrawal of consent, death and last safety follow-up visit (up to approximately 3 years)
  PFS is defined as time between the date of first dose of pembrolizumab and the date of either radiological disease progression, clinical/symptomatic disease progression or death (whichever is sooner).
Part C: Overall Survival (OS) | Baseline to death of any cause (up to approximately 3 years)
  OS is defined as time between the date of the first dose of study drug and the date of death due to any cause.
Part A2: Recurrence-free Survival (RFS) | Baseline up to 2 years
  RFS is defined as the time between the date of first dose of mRNA-4157 and the date of one of the following events: radiological disease relapse, clinical/symptomatic disease progression as assessed by the investigator or death due to any cause.
Parts A2, E1, E2, and E3: Number of Participants with Presence or Absence of Circulating Tumor DNA (ctDNA) | Baseline up to 2 years
  Presence or absence of ctDNA prior to start of treatment as well as across longitudinal study timepoints, and association with RFS.
Parts E1 and E2: Event-free Survival (EFS) | Baseline up to 2 years
  EFS is defined as the time from date of the first dose of study drug to the first of the following events: radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local, regional, or distant recurrence, or death due to any cause and will be determined either by biopsy assessed by local pathologist or by investigator-assessed imaging using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Part E3: EFS | Baseline up to 2 years
  EFS, based on RECIST 1.1, is defined as the time from date of the first dose of study drug to the first of the following events: radiographic disease progression per RECIST 1.1; local, regional or distant recurrence as assessed by computed tomography scan or biopsy if indicated (for participants who are disease free after surgery); clinical progression as evidenced by peritoneal carcinomatosis confirmed by preoperative laparoscopy or laparotomy (for participants who are confirmed to be free of peritoneal involvement by laparoscopy at screening); or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (8):
  - The George Washington Cancer Center, Washington D.C., District of Columbia
  - Orlando Health Cancer Institute, Orlando, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - NYU Langone Medical Center, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
- Australia (2):
  - Westmead Hospital-Cnr Hawkesbury and Darcy Road, Westmead, New South Wales
  - One Clinical Research Perth, Perth, Western Australia
- Japan (4):
  - National Cancer Center East, Chiba
  - Kindai University Hospital, Osaka
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Tokyo
- United Kingdom (3):
  - NHS Tayside, Dundee, Scotland
  - Royal Mardsen London, London
  - Royal Mardsen Sutton, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berraondo P, Cuesta R, Sanmamed MF, Melero I. Immunogenicity and Efficacy of Personalized Adjuvant mRNA Cancer Vaccines. Cancer Discov. 2024 Nov 1;14(11):2021-2024. doi: 10.1158/2159-8290.CD-24-1196. PMID 39485256